CLINICAL TRIAL: NCT02124486
Title: A Randomised Controlled Trial of Bariatric Surgery Versus a Community Weight Loss Programme for the Sustained Treatment of Idiopathic Intracranial Hypertension: the IIH:WT Trial
Brief Title: An RCT of Bariatric Surgery vs a Community Weight Loss Programme for the Sustained Treatment of IIH
Acronym: IIH:WT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr Alexandra Sinclair, NIHR Clinician Scientist and Honorary Consultant Neurologist, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_12-089; CS-011-028 (Other Grant/Funding Number: NIHR); 14/WM/0011 (Other: Black Country Research Ethics Committee); ISRCTN40152829 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: IIH; Weight loss; Bariatric surgery
MeSH Terms: conditions — Pseudotumor Cerebri; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dietetic Intervention (Active Comparator): Participants randomised to the dietetic arm will be given vouchers at baseline, 3, 6 and 9 months that exempt them from paying for consecutive and specified weeks of their local Weight Watchers diet programme.
  Interventions: Behavioral: Dietetic intervention
- Bariatric surgery (Experimental): Patients randomised to the bariatric surgery arm will be referred to the bariatric surgery pathway and, if judged suitable according to the bariatric surgery clinic's screening processes, undergo bariatric surgery.
  Interventions: Procedure: Bariatric surgery
- Matched obese control group (No Intervention): To evaluate the baseline difference in ICP between IIH patients and a matched obese control cohort we will recruit 20 obese but otherwise healthy participants who will undergo the same baseline visit as the main trial participants and then exit the study.
- MRI Test run (No Intervention): 5 patients will undergo double baseline MR scans to validate the novel MR sequences being used in the main trial.

INTERVENTIONS:
Procedure: Bariatric surgery — Participants randomised to the bariatric surgery arm of the trial will be referred to the surgery pathway according to NICE guidelines at Birmingham Heartlands Hospital (BHH), Heart of England NHS Foundation Trust.
  Arms: Bariatric surgery
Behavioral: Dietetic intervention — Participants randomised to the dietetic arm will be given vouchers at baseline, 3, 6 and 9 months that exempt them from paying for consecutive and specified weeks of their local Weight Watchers.
  Other Names: Weight Watchers
  Arms: Dietetic Intervention

SUMMARY:
Idiopathic intracranial hypertension (IIH) is a condition with an unknown cause or causes. The condition is associated with raised pressure in the brain and can cause disabling daily headaches and loss of sight, which can be permanent. The raised brain pressure squashes the nerves supplying the eye (also known as papilloedema) and this can affect vision. Over 90% of patients with IIH are overweight and weight loss is the most effective treatment. Other treatments for IIH have very little current evidence to support their use.

Weight loss is difficult to maintain. This trial aims to compare two methods of weight loss, bariatric surgery and the most effective dietary programme commonly available, Weight Watchers, to see which offers the most effective sustainable treatment for IIH. Bariatric surgery is recommended by the NICE clinical guidelines for patients with a Body Mass Index (BMI) of over 40, or over 35 with a co-morbidity. Women suffering from IIH have a BMI on average around 38 and IIH is not recognised as a co-morbidity for bariatric surgery.

This trial will recruit 64 women with IIH from Neurology and Ophthalmology clinics in UK NHS Trusts. They will be randomised and 32 participants will be allocated to the dietetic intervention arm, and be enrolled in their local Weight Watchers group. 32 participants will be allocated to the bariatric surgery arm, and will be referred to their local bariatric surgery pathway to receive bariatric surgery. Both groups of participants will be allocated to a treatment arm which is proven to bring about weight loss.

Participants will then be followed up for five years, with the most important measurement being their brain pressure after one year of being in the trial.

A further 20 obese women who don't suffer from IIH will be recruited to compare the baseline symptoms and biomarkers of those with IIH; they will take no further part in the study. 5 further healthy individuals will be scanned twice in an MRI test group to validate the MRI scan sequence to be used in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female IIH patients aged between 18 and 55 years, diagnosed according to the modified Dandy criteria who have chronic (> 6 months duration), active disease (papilloedema [Frisen grade ≥ 1], significantly raised ICP > 25cmH2O) and no evidence of venous sinus thrombosis (magnetic resonance or CT imaging and venography as noted at diagnosis).
2. BMI >35kg/m2.
3. Tried other appropriate non-surgical treatments to lose weight but have not been able to achieve or maintain adequate, clinically beneficial weight loss for at least 6 months.
4. Able to give informed consent.

Exclusion Criteria:

1. Age less than 18 or older than 55 years.
2. Pregnant or planning to conceive during the first 18 months of the trial .
3. Significant co-morbidity, endocrinopathy or the use of hormone manipulating medication (excluding contraception and topical or inhaled steroids).
4. Undergone optic nerve sheath fenestration.
5. Definite indication for or contraindication against surgery or dieting.
6. Have a specific medical or psychiatric contraindication for surgery, including drug misuse, eating disorder or major depression (suicidal ideation, drug overdose or psychological admission in last 12 months).
7. Previous bariatric surgery.
8. Taken AZD4017 within the last four months .
9. Inability to give informed consent e.g. due to cognitive impairment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-03-06 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
Intracranial Pressure | 12 months
  Change in Intracranial Pressure (ICP) between baseline and 12 months.
  ICP will be assessed using lumbar puncture (LP). To avoid the LP affecting the visual measures it will be performed after the visual tests have been completed. ICP will be recorded to the nearest whole number in cmH2O. Both opening and closing ICP will be recorded.

SECONDARY OUTCOMES:
Intracranial Pressure | 60 months
  Change in ICP between baseline and 24 and 60 months.
  ICP will be assessed using lumbar puncture (LP). To avoid the LP affecting the visual measures it will be performed after the visual tests have been completed. ICP will be recorded to the nearest whole number in cmH2O. Both opening and closing ICP will be recorded.
IIH symptoms | 12 months
  Change in reported IIH symptoms from 0 to 12 months (and at 3, 6, 24 and 60 months)
Visual function | 12 months
  Change in visual function from 0 to 12 months (and at 24 and 60 months).
  Assessments to be undertaken are the LogMAR (log of the minimum angle of resolution) chart to assess visual acuity, automated perimetry (Humphrey 24-2 central threshold) to measure the visual field mean deviation, an evaluation of contrast sensitivity and an Ishihara book to assess colour vision. The pupils will then be dilated using 1% tropicamide. Papilloedema will then be measured using spectral optical coherence tomography. Papilloedema will be further graded following fundus photographs. This will be done after all participants have reached the primary endpoint by two neuro-ophthalmologists blinded to trial treatment arm. The assessors will score the paired papilloedema images as better/same/worse as per the methodology described in a previous study. They will also assign a Frisen score to the images.
Papilloedema | 12 months
  Change in papilloedema from 0 to 12 months (and at 24 and 60 months)
Headache | 12 months
  Change in headache associated disability from 0 to 12 months (and at 24 and 60 months).
  Headache will be assessed by participant completed questionnaires. Participants will complete a daily headache diary in the week before assessments, which will evaluate the Headache Index score and use of analgesia (days/week). Headache associated disability will be evaluated using the Headache Impact Test-6 score (HIT 6). Severity and frequency of headaches will be assessed retrospectively using the Headache Index. Headache phenotype (according to criteria from the International Headache Society) will also be assessed.
Anthropometric measures | 12 months
  Change in anthropometric measures (e.g. waist, hip, fat mass) from 0 to 12 months (and at 24 and 60 months)
Quality of Life (EQ-5D-5L and SF-36) | 12 months
  Change in quality of life (participant reported) from 0 to 12 months (and at 24 and 60 months)
Referrals to CSF shunting procedures and optic nerve sheath fenestration | 12 months
  Difference in number of referrals to cerebrospinal fluid (CSF) shunting procedures and optic nerve sheath fenestration between treatment arms at 0 to 12 months (and at 24 and 60 months)
Health Economics | 12 months
  Health economics including cost-effectiveness at 12, 24 and 60 months.

OTHER OUTCOMES:
Biomarkers | 12 months
  Change in biomarkers from 0 to 12 (and 24 and 60) months
Matched control group comparison | Baseline
  Comparison between IIH patients and the matched control group at baseline with respect to biomarkers and ICP.
MRI Test Run | Baseline
  Change in MR imaging over a double baseline period of healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sinclair, MBChB, Principal Investigator — University of Birmingham
Locations (1):
- University Hospital Birmingham (Queen Elizabeth Hospital), Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Grech O, Seneviratne SY, Alimajstorovic Z, Yiangou A, Mitchell JL, Smith TB, Mollan SP, Lavery GG, Ludwig C, Sinclair AJ. Nuclear Magnetic Resonance Spectroscopy Metabolomics in Idiopathic Intracranial Hypertension to Identify Markers of Disease and Headache. Neurology. 2022 Oct 17;99(16):e1702-e1714. doi: 10.1212/WNL.0000000000201007. PMID 36240084
- [Derived] Mollan SP, Mitchell JL, Yiangou A, Ottridge RS, Alimajstorovic Z, Cartwright DM, Hickman SJ, Markey KA, Singhal R, Tahrani AA, Frew E, Brock K, Sinclair AJ. Association of Amount of Weight Lost After Bariatric Surgery With Intracranial Pressure in Women With Idiopathic Intracranial Hypertension. Neurology. 2022 Sep 13;99(11):e1090-e1099. doi: 10.1212/WNL.0000000000200839. Epub 2022 Jul 5. PMID 35790425
- [Derived] Mollan SP, Wakerley BR, Alimajstorovic Z, Mitchell J, Ottridge R, Yiangou A, Thaller M, Gupta A, Grech O, Lavery G, Brock K, Sinclair AJ. Intracranial pressure directly predicts headache morbidity in idiopathic intracranial hypertension. J Headache Pain. 2021 Oct 7;22(1):118. doi: 10.1186/s10194-021-01321-8. PMID 34620087
- [Derived] Yiangou A, Mitchell JL, Nicholls M, Chong YJ, Vijay V, Wakerley BR, Lavery GG, Tahrani AA, Mollan SP, Sinclair AJ. Obstructive sleep apnoea in women with idiopathic intracranial hypertension: a sub-study of the idiopathic intracranial hypertension weight randomised controlled trial (IIH: WT). J Neurol. 2022 Apr;269(4):1945-1956. doi: 10.1007/s00415-021-10700-9. Epub 2021 Aug 22. PMID 34420064
- [Derived] Mollan SP, Mitchell JL, Ottridge RS, Aguiar M, Yiangou A, Alimajstorovic Z, Cartwright DM, Grech O, Lavery GG, Westgate CSJ, Vijay V, Scotton W, Wakerley BR, Matthews TD, Ansons A, Hickman SJ, Benzimra J, Rick C, Singhal R, Tahrani AA, Brock K, Frew E, Sinclair AJ. Effectiveness of Bariatric Surgery vs Community Weight Management Intervention for the Treatment of Idiopathic Intracranial Hypertension: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):678-686. doi: 10.1001/jamaneurol.2021.0659. PMID 33900360
- [Derived] Ottridge R, Mollan SP, Botfield H, Frew E, Ives NJ, Matthews T, Mitchell J, Rick C, Singhal R, Woolley R, Sinclair AJ. Randomised controlled trial of bariatric surgery versus a community weight loss programme for the sustained treatment of idiopathic intracranial hypertension: the Idiopathic Intracranial Hypertension Weight Trial (IIH:WT) protocol. BMJ Open. 2017 Sep 27;7(9):e017426. doi: 10.1136/bmjopen-2017-017426. PMID 28963303